CLINICAL TRIAL: NCT03325127
Title: Outcomes and Treatment Patterns of Metastatic Castration Resistant Prostate Cancer (mCRPC) Patients Treated With Radium-223 Concomitantly With Abiraterone or Enzalutamide in First Line Setting : A Retrospective Chart Abstraction Study
Brief Title: Outcomes of mCRPC Patients Treated With Ra-223 Concomitant With Abiraterone or Enzalutamide- A Chart Review Study
Status: Withdrawn | Type: Observational
Why Stopped: Project plan changed, study conduct was no longer needed.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19706
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: Prostate Cancer, Bone metastases, Xofigo, Zytiga, Xtandi.
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms | interventions — radium Ra 223 dichloride; Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radium-223 concomitant with Abiraterone or Enzalutamide: Approximately 150 medical charts from mCRPC patients within the network will be collected
  Interventions: Drug: radium Ra 223 dichloride (Xofigo, BAY88-8223); Drug: Zytiga; Drug: Xtandi

INTERVENTIONS:
Drug: radium Ra 223 dichloride (Xofigo, BAY88-8223) — Radium-223, 55kBq (1.49 microcurie) per kg body weight given at 4 week intervals for 6 injections
Drug: Zytiga — Abiraterone 1000 mg per day orally
Drug: Xtandi — Enzalutamide 160 mg per day orally

SUMMARY:
There are no real-world data that describes how Radium-223 (Ra-223) is being used in combination with abiraterone/enzalutamide (abi/enza) or evidence describing outcomes of this combination usage for the treatment of metastatic castration resistant prostate cancer (mCRPC). To address these data gaps a cohort of mCRPC patients will be chosen who received Ra-223 concomitant with abi/enza in first line therapy to assess the treatment patterns following first line and clinical outcomes from initiation of first line treatment. For the purpose of this study concomitant use will be defined as Ra-223 initiated after at least 6 months from the start of first line abi/enza. The specific objectives of the study are to describe the outcomes, treatment patterns, patient and provider characteristics of mCRPC patients treated with Ra-223 concomittantly with abi/enza in first line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mCRPC and bone metastases
* ≥ 40 years of age at diagnosis of mCRPC
* Initiated first line treatment for mCRPC with abi/enza (use of sipuleucel-T prior to initiation of abi or enza is allowed)
* Receipt of at least one cycle of radium-223 after 15 May 2013
* First cycle of Ra-223 occurs while receiving first line treatment with abi/enza
* Treated with abi/enza for at least 28 days (1 cycle) following initiation of Ra-223
* Initiation of Ra-223 at least 6 months after the start of treatment with abi/enza
* Completion of Ra-223 treatment prior to the receipt of any chemotherapy for mCRPC
* At least 12 months of follow-up (or until death) from date of initiation of Ra-223
* Known date of death (if patient deceased)

Exclusion Criteria:

* Receipt of any prior chemotherapy during hormone sensitive disease or any time before mCPRC
* Active participant in an interventional clinical trial for CRPC in first line
* Presence of visceral metastases at initiation of Ra-223 treatment
* Treated with abi/enza (with or without docetaxel) prior to the development of metastatic and/or castration resistant disease

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by their treating physicians (oncologists and urologists), who will be recruited for participation in the research from the Cardinal Health Oncology Research Network (CHORN).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10-30 (Estimated); Primary Completion 2018-09-28 (Estimated); Study Completion 2018-09-28 (Estimated)

PRIMARY OUTCOMES:
Survival rates | Up to 1 year
  Survival will be defined as time from initiation of first line therapy until death. Survival will be measured as the proportion of study subjects that are alive at the data cut-off or median time for survival of at least 50% of study subjects

SECONDARY OUTCOMES:
Disease progression | Up to 1 year
  Disease progression will be defined as either of the below:
  PSA (Prostate Specific Antigen) progression ALP (Alkaline Phosphatase) progression Symptomatic progression Radiographic progression
Skeletal related events (SRE) | Up to 1 year
  SRE will be defined as: a pathologic fracture, spinal cord compression, necessity for radiation to bone for pain or impending fracture and/or surgery to bone
Symptomatic Skeletal Events (SSE) | Up to 1 year
  SSE defined as external beam radiation therapy (EBRT) to relieve skeletal symptoms, new symptomatic pathologic bone fracture, occurrence of spinal cord compression, or tumor-related orthopedic surgical intervention
Time to death | Up to 1 year
Sequence of treatment regimens | Up to 1 year
Dose schedule | Up to 1 year
Duration of therapy | Up to 1 year
Time to first visceral metastasis | Up to 1 year
Proportion of patients developing visceral metastasis | Up to 1 year